

<Protocol: Janssen OZ1-HV1-101/102/202>

<INC code: 1003733> <SAP Version: 3.0>

PROJECT MANAGER:

#### STATISTICAL ANALYSIS PLAN

INC STUDY NO.: 1003733

AUTHOR:

DATE OF ISSUE: Nov 7th, 2017

SPONSOR: Janssen Cilag

STUDY TITLE: Long term follow-up of the following:

A marker study of therapeutically transduced CD4+ peripheral blood lymphocytes in HIV discordant

identical twins (Protocol OZ1-HV1-101)

A Phase I trial of autologous CD34+ hematopoietic

progenitor cells transduced with an anti-HIV

ribozyme (Protocol OZ1-HV1-102)

A long term follow-up protocol to evaluate the

safety and survival of autologous CD34+

hematopoietic progenitor cells transduced with an anti-HIV-1 ribozyme (OZ1) in patients with HIV-1 infection (*Protocol OZ1-HV1-202 Amendment 4*)



<Protocol: Janssen OZ1-HV1-101/102/202>

<INC code: 1003733> < SAP Version: 3.0>

### **Signature Page**

Version: Final 3.0

Version Date: Nov 7th, 2017

I confirm that I have reviewed this document and agree with the content.

| Designation | Print Name | Signature | Date |
|---|---|---|---|
| Sponsor<br>Representative | | | Date 20 8.01.02 16:37:49 +08:00* |
| Lead Statistician | | | 20-PEC-2017 |
| Lead Statistical<br>Programmer | | | 2200(2017 |
| Project Manager | | | 22 Dec 2017 |



<Protocol: Janssen OZ1-HV1-101/102/202>


### **TABLE OF CONTENTS**

| 1. | INTRODUCTION | 6 |
|------|------------------------------------------------|----|
| 1.1. | Responsibilities | 6 |
| 1.2. | Glossary of Abbreviations | 7 |
| 1.3. | Defintion of Terms | 8 |
| 2. | OBJECTIVES | 9 |
| 3. | STUDY DESIGN | 10 |
| 3.1. | Overview of Study Design | 10 |
| 3.2. | Study Sample Size | 12 |
| 4. | POPULATIONS FOR ANALYSIS | 13 |
| 4.1. | Safety Population | 13 |
| 4.2. | Per-Protocol Population | 13 |
| 5. | OVERALL CONSIDERATIONS | 14 |
| 6. | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | 15 |
| 6.1. | Demographic Characteristics | 15 |
| 6.2. | Patient Disposition and Withdrawals | 15 |
| 6.3. | Significant Medical History | 16 |
| 6.4. | Other Initial Study Information | 16 |
| 7. | <u>EFFICACY</u> | 18 |
| 7.1. | Marking in Peripheral Blood Mononuclear Cells | 18 |



| <protocol:< th=""><th>Janssen</th><th>OZ1-HV1</th><th>-101/</th><th>102/202&gt;</th></protocol:<> | Janssen | OZ1-HV1 | -101/ | 102/202> |
|---|---|---|---|---|
|---|---|---|---|---|


| <b>7.2.</b><br>7.2 | | |
|---|---|---|
| 8. <u>s</u> | SAFETY | .20 |
| 8.1. | Compliance | 20 |
| 8.2 | .2. Summary of SAÉs by System Organ Class, Preferred Term, Severity and ationship | 21 |
| 8.2<br>8.2 | , , | |
| 8.3. | Predominant Integration Site Test | 23 |
| 8.4. | CBC/Differential and Platelets | 23 |
| 8.5. | Clinical History | 23 |
| 8.6. | Replication Competent Retrovirus | 24 |
| 8.7. | Physical Examination | 24 |
| 9. <u>I</u> | NTERIM ANALYSES | . 25 |
| 10.<br><u>ANA</u> | CHANGES IN THE CONDUCT OF THE STUDY OR PLANNNED LYSIS | .26 |
| 10.1. | Changes in the Conduct of the Study | 26 |
| 10.2. | Changes to the Analyses Planned in the Study | 26 |
| 11. | REFERENCE LIST | .27 |
| 12. | PROGRAMMING CONVENTIONS | . 28 |
| 13. | INDEX OF TABLES | .29 |



| <protocol:< th=""><th>lanssen</th><th>071-HV1</th><th>-101/</th><th>/102/202&gt;</th></protocol:<> | lanssen | 071-HV1 | -101/ | /102/202> |
|---|---|---|---|---|


| 14. | INDEX OF FIGURES | 31 |
|-----|-------------------|----|
| 15. | INDEX OF LISTINGS | 32 |



<Protocol: Janssen OZ1-HV1-101/102/202>


### 1. <u>INTRODUCTION</u>

#### 1.1. RESPONSIBILITIES

This document details the proposed tabular and graphical presentations of data collected from long term cell delivered rybozyme gene transfer product (OZ1) follow up studies; OZ1-HV1-101, OZ1-HV1-102 and OZ1-HV1-202. This document also defines the analysis populations and the safety and efficacy endpoints.

This document has been written by INC based on information contained in the study protocols OZ1-HV1-101 amendment 2 dated 23 October 2007, OZ1-HV1-102 amendment 2 dated 23 October 2007, and OZ1-HV1-202 amendment 2 dated 28 August 2007 and OZ1-HV1-202 amendment 4 dated 07 Jun 2017

The production of summary tables, data listings, graphs and statistical analyses will be the responsibility of Biometrics at INC, and will be performed according to INC standard operating procedures (SOPs).

One completed analysis which was reported in 2011 covered data collected from the point of First Patient First Visit (FPFV) in January 2000 until the last subject year 5 follow-up visit (Last Patient Last Visit: LPLV) in February 2011. A separate Statistical Analysis Plan (SAP) was used for this previous analysis (Kendle study 76803). This previous SAP has also been used as a template for this new INC study (1003733).

This SAP had covered an interim analysis in 2016 and will cover a final analysis happened after DBL of study *OZ1-HV1-202*. The interim analysis in 2016 was based on cumulative data collected from the point of First Patient First Visit (FPFV) in January 2000 until the last subject year 10 follow-up visit (Last Patient Last Visit (LPLV) in February 2016. The final analysis expected in 2018 will be based on cumulative data collected from the point of FPFV in January 2000 until the last subject completes the end of study visit by 30-Nov-2017.

The previous Kendle study (76803) database used TrialBase software and the new INC study (1003733) database will use Oracle Clinical software. Data extracts from each database into SAS will be combined to create analysis datasets covering the cumulative data from both databases. The analyses in 2018 covered in this SAP will also be based on clean data.



<Protocol: Janssen OZ1-HV1-101/102/202>


#### 1.2. GLOSSARY OF ABBREVIATIONS

AE Adverse event

CBC Complete blood count CD Cluster of differentiation

CRF Case report form

FDA United States Food and Drug

Administration

FPFV First Patient First Visit

HIV Human immunodeficiency virus

LNL6 Moloney murine leukemia virus based

retroviral vector

LPLV Last Patient Last Visit

MedDRA Medical Dictionary for Regulatory Activities

n Number of observations

NSRAE Non-serious related adverse events

OZ1 Cell delivered rybozyme gene transfer

product

PBMC Peripheral blood mononuclear cells

PCR Polymerase chain reaction RCR Replication competent retrovirus

SAE Serious adverse event SAP Statistical Analysis Plan

SOP Standard operating procedure



<Protocol: Janssen OZ1-HV1-101/102/202>


#### 1.3. DEFINTION OF TERMS

The following terms will be used throughout this statistical analysis plan to refer to the three contributing protocols.

| 101 | OZ1-HV1-101 long term follow-up |
|-----|---------------------------------|
| 102 | OZ1-HV1-102 long term follow-up |
| 202 | OZ1-HV1-202 long term follow-up |

The phrase 'long term follow-up' used throughout this SAP refers to each individual long term follow-up of 101, 102 and 202.

For the purposes of this SAP the term 'adverse events' refers to all serious and non-serious related adverse events only.

All subject ID numbers consist of 6 characters. The following subject ID applies to each of the protocols.

| 101 | 0R000X |
|-----|--------|
| 102 | 0000XX |
| 202 | OZ1XXX |

Where X represent the individual subject number.

Research\*

<Protocol: Janssen OZ1-HV1-101/102/202>


### 2. OBJECTIVES

- 1. To undertake long term safety monitoring for any development of:
  - a. Clonal expansion of cells with a predominant OZ1 (or LNL6 vector) insertion site
  - b. Insertional oncogenesis
- 2. To archive/store plasma and peripheral blood mononuclear cells (PBMC) samples for other safety testing that may be required.
- 3. To assess quantitative marking of the gene transfer product in PBMCs over time. The 202 protocol includes the assessment of quantitative marking and expression of the gene transfer product in PBMCs over time.



<Protocol: Janssen OZ1-HV1-101/102/202>


### 3. <u>STUDY DESIGN</u>

#### 3.1. OVERVIEW OF STUDY DESIGN

The OZ1-HV1-101, OZ1-HV1-102 and OZ1-HV1-202 studies form the long term follow-up for OZ1. OZ1 comprises a Moloney Murine Leukemia Virus based retroviral vector (LNL6) containing a gene that encodes an anti-human immunodeficiency virus (HIV) ribozyme. It is a recommendation of the United States Food and Drug Administration (FDA) that all individuals receiving retroviral gene transfer products are followed for life.

Patients who participated in the Phase I study "A Marker Study of Therapeutically Transduced CD4+ Peripheral Blood Lymphocytes in HIV discordant twins" were asked to continue long term monitoring under the OZ1-HV1-101 protocol. Patients who participated in the Phase I study "A Phase I Trial of Autologous CD34+ Hematopoietic Progenitor Cells Transduced with an Anti-HIV Ribozyme" were to continued long term monitoring under the OZ1-HV1-102 protocol. Patients who participated in the Phase II study "A randomized Phase II, double blind, controlled trial to evaluate the safety and efficacy of autologous CD34+ hematopoietic progenitor cells transduced with placebo or an anti-HIV ribozyme (OZ1) in patients with HIV-1 infection" continue long term monitoring under the OZ1-HV1-202 protocol. Following completion and unblinding of the Phase II study, patients who were identified as having been enrolled in the placebo arm were subsequently discontinued from the long term follow-up study 202.

All patients in each protocol will be reviewed at 6 month intervals (+/- 6 weeks) until year 5 post infusion. Thereafter, all patients will be reviewed annually (+/- 12 weeks) on the anniversary of their infusion. Given the recommendation to follow patients for life, patients who withdraw from the study or have been lost to follow-up but return for assessments at a later time may be re-instated in their study. Additional unscheduled visits may be made if any clinical or biological findings require further investigation. A schedule detailing the timing of the follow-up visits and the procedures carried out at each visit is presented in Table 1.

Various data and samples have been collected under previous protocol versions. For data consistency across all the long term follow-up protocols only data corresponding to the schedule presented in Table 1 collected on one standardized Case Report Form (CRF) will be included in the data analysis. Additionally, the CRF will collect 'Initial Study Information' which will comprise of demography, significant medical history, treatment details from the respective original studies, and PBMC analysis and complete blood count (CBC)/differential and platelets results obtained 2 years post infusion or the nearest timepoint before starting the respective long term follow-up if 2 years post infusion data is not available.




<Protocol: Janssen OZ1-HV1-101/102/202>


#### Table 1 Visit Schedule

| Follow-up Visit | | Year | Year | Year | Year | Annual Visit | Annual Visit<br>Year 15+ |
|---|---|---|---|---|---|---|---|
| | 2.5 | 3 | 3.5 | 4 | 4.5 | Year 5-15 | real 15+ |
| Clinical history and examination | X | X | X | Χ | X | X | X |
| Complete Blood Count (CBC)/Differential and Platelets | Χ | Χ | Χ | Χ | Χ | X | |
| Plasma archive | | Χ | | Χ | | X | X |
| PBMC archive <sup>1</sup> | | X | | Χ | | X | X |
| OZ1 integration site polymerase chain reaction (PCR) <sup>2</sup> | | Х | Х | Х | Х | X | |
| Adverse Events Assessments | | Χ | Χ | Χ | Χ | X | X |
| Contact details updated for patient and nominated secondary contact | | Х | Х | Х | Х | X | X |

<sup>&</sup>lt;sup>1</sup>The PBMCs will be stored as cryopreserved cells and cell pellets for replication competent retrovirus (RCR) and other safety testing as required.

<sup>2</sup>This includes both marking (quantitative OZ1/LNL6 DNA-PCR) and the detection of predominant integration sites. If the percentage of cells marked by the vector (quantitative OZ1/LNL6 DNA-PCR) is less than 1% of the test cell population, the site of integration will not be investigated. If a predominant integration site is detected, the patient will be retested within 3 months to determine if it persists. If so, the site of integration of OZ1 will be sequenced and mapped to the human genome to determine any association with known human oncogene. In all instances that a predominant integration site is present and, particularly when there is expansion of a cellular clone, the patient will be monitored for signs of cancer, so that treatment can be initiated as early as possible. Ongoing analysis of quantitative marking of the gene transfer product will be performed as part of the testing of predominant integration sites. These marking data will also be analyzed independently to detect any changes in the number of cells carrying the gene transfer product.

<sup>3</sup>Blood can be collected up to 1 week prior to the other assessments.



<Protocol: Janssen OZ1-HV1-101/102/202>


#### Table 2 Visit Schedule (Study 202)

| | | | | | | Annual |
|---|---|---|---|---|---|---|
| Follow up visit | Yr 2.5 | Yr 3 | Yr 3.5 | Yr 4 | Yr 4.5 | Yr 5+<br>/End-of-Study <sup>4</sup> |
| Clinical history and examination | X | X | X | X | X | X |
| Complete Blood Count/Differential and Platelets | X | X | X | X | X | X |
| Plasma archive | | X | | X | | X |
| PBMC archive <sup>1</sup> | | X | | X | | X |
| OZ1 integration site (PCR) <sup>2</sup> | X | X | X | X | X | X |
| Adverse Events Assessment | X | X | X | X | X | X |
| Contact details updated for subject and nominated secondary contact | X | X | X | X | X | X |
| Volume of blood drawn at visit (ml) <sup>3</sup> | 30 | 73 | 30 | 73 | 30 | 73 |

<sup>&</sup>lt;sup>1</sup>The PBMCs will be stored as cryopreserved cells and cell pellets for assessment of replication competent retrovirus (RCR) and other safety testing as required.



<Protocol: Janssen OZ1-HV1-101/102/202>


<sup>2</sup>This includes both marking (quantitative OZ1/LNL6 DNA-PCR) and the detection of predominant integration sites. If the percentage of cells marked by the vector (quantitative OZ1/LNL6 DNA-PCR) is less than 1% of the test cell population, the site of integration will not be investigated. If a predominant OZ1 integration site is detected, the patient will be retested within 3 months to determine if it persists. If so, the site of integration of OZ1 will be sequenced and mapped to the human genome to determine any association with a known human oncogene. In all instances that a predominant integration site is present and, particularly when there is expansion of a cellular clone, the patient will be monitored for signs of cancer, so that treatment can be initiated as early as possible. Ongoing analysis of quantitative marking of the gene transfer product will be performed as part of the testing of predominant integration sites. These marking data will also be analyzed independently to detect any changes in the number of cells carrying the gene transfer product.

<sup>3</sup>Blood can be collected up to 1 week prior to the other assessments.

<sup>&</sup>lt;sup>4</sup> End-of-Study assessments will be performed after all ongoing patients have been followed up for least 10 years post-infusion. End-of-Study visits will be completed by 30 November 2017. In the event that a patient cannot attend a site visit, telephonic follow-up will be an acceptable alternative.

Research®

<Protocol: Janssen OZ1-HV1-101/102/202>


#### 3.2. STUDY SAMPLE SIZE

The sample size of the long term follow-up studies is dependant on the number of patients continuing into the long term follow-up phase from the original studies. No formal sample size calculation was performed.



<Protocol: Janssen OZ1-HV1-101/102/202>


### 4. **POPULATIONS FOR ANALYSIS**

Assignment of patients to each of the populations together with a review of the data will take place at a Data Review Meeting to be held immediately prior to database lock. All decisions taken at the Data Review Meeting regarding the analysis populations will be fully documented.

The following listings will be provided for the Data Review Meeting:

Demography (Listing 16.2.2)
Significant Medical History (Listing 16.2.3)
Treatment Details (Listing 16.2.4)

PBMC Analysis (Listings 16.2.5.1, 16.2.5.2, 16.2.5.3)

Patient Disposition (Listing 16.2.1.1)
Clinical History (Listing 16.2.12)
Discontinuation Details (Listing 16.2.1.2)
Re-instatement Details (Listing 16.2.1.3)

Adverse Events (Listings 16.2.8.2, 16.2.8.3)

Death (Listing 16.2.8.1)

Proposed analysis Populations

together with reasons for exclusion (Listing 16.2.1.4)

Other listings may be provided for the Data Review Meeting as required.

#### 4.1. SAFETY POPULATION

The Safety population will consist of any patient who was enrolled in either of the OZ1-HV1-101, OZ1-HV1-102 or OZ1-HV1-202 studies and continued into the respective long term follow-up protocol.

#### 4.2. PER-PROTOCOL POPULATION

All patients who are eligible for inclusion in the Safety population and received OZ1 or LNL6 or combination OZ1/LNL6.



<Protocol: Janssen OZ1-HV1-101/102/202>


#### 5. OVERALL CONSIDERATIONS

All summary tables and data listings produced by INC will use the statistical package SAS (v9.2 or a more recent version).

In general, categorical data will be presented using counts and percentages, whilst continuous data will be presented using the descriptive statistics, mean, standard deviation (SD), median, minimum, maximum and number of patients with an observation (n). Minimum and maximum values will be quoted to the number of decimal places as recorded on the CRF; means, medians and SDs will be quoted to one further decimal place. Percentages will be rounded to one decimal place. Percentages smaller than 0.1 will be presented as <0.1. Percentages whose numerator is zero will be reported as zero.

All data recorded on the Case Report Form (CRF) and any derived data will be listed for all patients.

The Safety population will be used to present Adverse Event and death data. The PP population will be used to present all data .

Unless otherwise stated missing data will not be imputed. Patients who withdraw prematurely will have their data summarized at the last attended visit. Repeat assessments will not be summarized unless otherwise indicated but will be fully listed. Similarly, data collected at unscheduled visits will be listed only. Repeat and unscheduled visits will be identified on the data listings.

Where of interest, presentation of data will be pooled to reflect the target cell type, CD4 cells in OZ1-HV1-101 and CD34 cells in OZ1-HV1-102 and OZ1-HV1-202 in addition to presenting separately and overall.

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


# 6. <u>DEMOGRAPHIC AND OTHER BASELINE</u> <u>CHARACTERISTICS</u>

#### 6.1. DEMOGRAPHIC CHARACTERISTICS

Date of birth, gender and race are recorded on the CRF as part of the initial study information.

Age (years) will be calculated using the formulae below and rounded to 1 decimal place.

Age at Infusion = (Date of Infusion - Date of Birth) / 365.25 Age at Database Lock Cut Off = (Date of cut off\* - Date of Birth) / 365.25

\* According to the current patient visit schedule this is due 13FEB2016 (window period +/-6 weeks). If a patient has discontinued or died before the date of cut off, the date of Study Discontinuation will replace date of cut off.

Age will be summarized using descriptive statistics, mean, median, standard deviation (SD), minimum, maximum and n separately for patients in 101, 102, 202 and overall.

The number and percentage of patients within each category for gender and race will be summarized for patients in 101, 102, 202 and overall.

Demography will be summarized for PP population.

#### 6.2. PATIENT DISPOSITION AND WITHDRAWALS

The number and percentage of patients who are ongoing and have never discontinued, discontinued and re-instated, and discontinued and never re-instated will be presented separately for 101, 102, 202 and overall. The primary reason for withdrawal will also be presented for those patients who have discontinued.

A table detailing the visit and date of last visit prior to discontinuation together with the reason for discontinuation of each individual patient who discontinued during the long term follow-up will also be presented.

Patients may be discontinued from the long term follow-up for any of the following reasons:

- Patient request
- Were randomized to the placebo treatment arm (202 only)



<Protocol: Janssen OZ1-HV1-101/102/202>


- Lost to follow-up
- Regulatory authority request
- Study termination
- Other

Patient disposition and withdrawal data will be summarized for all patients.

The number and percentage of patients assigned to each analysis population will be summarized separately for 101, 102 and 202 and overall.

#### 6.3. SIGNIFICANT MEDICAL HISTORY

Information relating specifically to HIV-1 infection will be recorded in the significant medical history (body system Immunological/Rheumatological) as part of the initial study information.

Time since HIV-1 infection will be summarized by descriptive statistics, mean, median, standard deviation (SD), minimum, maximum and n separately for 101, 102 and 202 and overall for the Safety and PP populations. Time since HIV-1 infection will be derived as follows:

Time since HIV-1 infection (yrs) = Year of diagnosis – (Date of Database lock + 1)

Data recorded for other body systems will be listed only.

#### 6.4. OTHER INITIAL STUDY INFORMATION

Treatment details (date of infusion, dose, treatment and transduced efficiency) from the original studies are recorded as part of the initial study information. Patients in 101 originally received a single dose of transduced CD4+ lymphocytes and patients in 102 and 202 originally received a single dose of CD34+ cells.

Time since infusion (years) will be derived using the following formula:

(Date of Last Visit in Long Term Follow-up – Date of Infusion) / 365.25

Time since infusion, dose, transduction efficiency and calculated dose will be summarized using descriptive statistics, mean, median, standard deviation, minimum, maximum and n by cell type (CD4 or CD34). Calculated dose will be derived as follows:

Dose (CD4+ or CD34+) / 100 x transduction efficiency



<Protocol: Janssen OZ1-HV1-101/102/202>


#### 7. EFFICACY

#### 7.1. MARKING IN PERIPHERAL BLOOD MONONUCLEAR CELLS

PBMC analysis (OZ1 & LNL6 DNA PCR (marking)) will be performed at 2 years post infusion or the nearest timepoint before starting the long term follow-up and at each 6 monthly visit up to 5 years post infusion and annually there after. Analyzed samples for gene detection will be classified as either not done, not detected or detected. If detected genes are found these will further be classified as to whether they are below the limit of quantification or not. Samples below the limit of quantification will be classified as either 1/3 (genes detected in 1 of the 3 triplicates of the sample), 2/3 (genes detected in 2 of the 3 triplicates of the sample) or 3/3 (genes detected in 3 of the 3 triplicates of the sample). For samples above the limit of quantification the percentage detected will be recorded for OZ1 & LNL6 DNA-PCR.

#### 7.2. METHODS OF ANALYSIS

#### 7.2.1. Analysis of Marking in Peripheral Blood Mononuclear Cells

For OZ1 & LNL6 DNA-PCR (marking) the number and percentage of patients in each of the categories Not Detected, Detected (1/3 Detected, 2/3 Detected, 3/3 Detected) and Detected (Quantifiable). The number and percentage of patients in each category will be presented at each timepoint for 102/202 combined and overall for the PP population.

Patients who have quantifiable OZ1 & LNL6 DNA-PCR detected will have the value listed and the relationship between the % marking and calculated dose, age at infusion, gender and race explored as described below.

Correlation between OZ1 & LNL6 DNA-PCR (%) and calculated dose will be assessed using PROC CORR in SAS. The number of patients with quantifiable detected and calculated dose data, Spearman's rank correlation co-efficient and its associated p-value will be presented. Similar presentations will be made for OZ1 & LNL6 DNA-PCR (%) versus age and OZ1 & LNL6 DNA-PCR (%) and time since infusion (as defined in Section 6.3).

Association between the number of patients with and without OZ1 & LNL6 DNA-PCR quantifiable detection and gender will be assessed by the Chi-Squared test using PROC FREQ in SAS. The number of patients with data for both parameters, the Chi-Square statistic and its associated p-value will be presented. A p-value of less than 0.05 will indicate an association between the parameters. Similar presentations will be made for OZ1 & LNL6 DNA-PCR versus race and gender. If it is not appropriate to perform the Chi-Square test due to small cell sizes, Fishers Exact test will be performed.

Research®

<Protocol: Janssen OZ1-HV1-101/102/202>


The above analyses will be performed for 102/202 combined and overall at each post infusion timepoint for the PP population providing there are patients with quantifiable data to render the analyses meaningful. A review of the marker data will take place at the Data Review Meeting. All decisions taken regarding the above analyses will be fully documented in the meeting minutes.

The percentage of patients detected with either a quantifiable or non quantifiable OZ1 & LNL6 DNA-PCR result will be plotted over time for 101, 102 and 202 separately, 102/202 combined and overall for the PP population.

Research®

<Protocol: Janssen OZ1-HV1-101/102/202>


#### 8. <u>SAFETY</u>

#### 8.1. COMPLIANCE

Patient compliance to visit attendance will be calculated using the following formula:

Number of Visits Eligible to Attend – Number of Eligible Visits Not Attended x 100

Number of Visits Eligible to Attend

Where the number of visits eligible to attend will be derived for each patient from the time of infusion *i.e.* 5 years since infusion = 6 visits in long term follow-up at 2.5, 3, 3.5, 4, 4.5 and 5 years, etc. Repeat or unscheduled visits will not be included in the above calculation.

Visit compliance will be summarized using descriptive statistics, mean, median, standard deviation (SD), minimum, maximum and n separately by time since infusion (≤ 5 yrs, > 5 yrs/≤10yrs and >10yrs) for 101, 102 and 202 and overall for PP population.

#### 8.2. ADVERSE EVENTS

Throughout the long term follow-up, all serious adverse events (SAEs) and non-serious related adverse events (NSRAEs) observed by medical staff, or reported by the patient, will be evaluated by the investigator and noted in the adverse event section of the CRF.

SAEs and NSRAEs will be coded using the current Medical Dictionary for Regulatory Activities (MedDRA). SAEs and NSRAEs will be summarized separately for 101, 102 and 202 and overall by tabulating the frequency of reports for each unique event and by tabulating the number of patients experiencing one or more events. The denominator used for the calculation of percentages will be the number of patients in the Safety population for the respective long term follow-ups. SAEs and NSRAEs will be summarized by MedDRA system order class and preferred term. Separate data listings of all information relating to patient death, SAEs and NSRAEs will be provided.

SAEs are defined as events that have a seriousness category of death, life threatening, initial or prolonged hospitalization, disability, congenital anomaly or other medically important condition such as predominant integration site, positive RCR, malignancy or abnormal pregnancy outcome (*ie* recorded seriousness category of 1, 2, 3, 4, 5 or 6). AEs recorded as non-serious (7) will be defined as non-serious and will only be recorded if they are considered related to the gene transfer product. A related AE is defined as any



<Protocol: Janssen OZ1-HV1-101/102/202>


AE whose relationship to the gene transfer product is recorded as possible, probable or very likely (coded on CRF as 3, 4, or 5). Severe AEs are defined as any AE recorded in the 'severe' category (coded on CRF as 3). AEs leading to death are defined as any AE in the seriousness category of 'death' (coded on CRF as 1) and/or an outcome category of 'fatal' (coded on CRF as 5). NSRAEs are defined as adverse events (AEs) whose seriousness category is recorded as non-serious but are considered to have a possible, probable or very likely relationship to the gene transfer product.

If the severity or relationship of an SAE/AE is missing a worst case scenario will be assumed (*ie* the AE will be set to severe or very likely, respectively).

The following AE summary tables will be presented 101, 102, 202 and overall.

#### 8.2.1. Overall Summary of Adverse Events

The following will be summarized:

Number and percentage of patients with at least one SAE
Number and percentage of patients with at least one related SAE
Number and percentage of patients with at least one severe, related SAE
Number and percentage of patients with at least one NSRAEs
Number and percentage of patients with SAE leading to death

Number of SAEs Number of related SAEs Number of severe related SAEs Number of NSRAEs Number of SAE/NSRAE leading to death

## 8.2.2. Summary of SAEs by System Organ Class, Preferred Term, Severity and Relationship

SAEs will be tabulated (n and %) within each severity category (mild, moderate, severe) and overall categories by system organ class and preferred term. In addition, the number of SAEs will be presented by relationship. Related SAEs are defined as those events coded as 'possible', 'probable' or 'very likely'. Non related SAEs are defined as those events coded as not related or doubtful. Counts will be given for both system organ class and preferred term. Each patient experiencing an SAE will be identified within preferred term and shown under the maximum severity relating to the particular preferred term. For overall severity categories, relationship of the AE will take priority over severity *ie* for the same patient a mild related headache will be counted over an unrelated severe headache.



<Protocol: Janssen OZ1-HV1-101/102/202>


For both system organ class and preferred term, counting will be done by patient and not by event. A patient will only be counted once within each system organ class and preferred term. The maximum severity for an event will be taken for each patient.

## 8.2.3. Summary of SAEs and Non-Serious Related Adverse Events by System Organ Class, Preferred Term, Outcome and Relationship

SAEs and NSRAEs will be tabulated (n and %) within each outcome category (recovered/resolved, recovering/resolving, not recovered/not resolved, recovered with sequelae, fatal, unknown) by system organ class, preferred term. In addition, the number of SAEs and NSRAEs will be presented by relationship. Related SAEs are defined as those events coded as possible, probable or very likely. Not related SAEs are defined as those events coded as not related or doubtful. Counts will be given for both system organ class and preferred term. Each patient experiencing a related SAE will be identified within preferred term and shown under the outcome relating to the particular preferred term.

For both system organ class and preferred term, counting will be done by patient and not by event. A patient will only be counted once within each system organ class and preferred term.

## 8.2.4. Summary of Time Adjusted Related SAEs by System Organ Class and Preferred Term

The number of related SAEs will be presented by system organ class and preferred term. In addition, event rate per year will be calculated using the formula below:

Event rate per year = Number of related SAEs / Patient years in long term follow-up

Where patient years in long term follow-up is calculated individually for each patient using the last available date of a safety assessment – (date of infusion + 2 yrs) and summed over all patients.

Each value from the above derivation will be totaled over each body system and preferred term to give a rate at which a particular related SAE may be experienced by a patient in a given year *ie* a patient rate per year of 1 for a particular preferred term is equal to a patient experiencing a related SAE once a year for the particular preferred term.

## 8.2.5. Correlation between Frequency of SAEs and NSRAE and Time on Study

Correlation between OZ1 & LNL6 DNA-PCR (%) and the frequency of SAEs and NSRAEs will be assessed using PROC CORR in SAS. The number of patients on study and experiencing at least one SAE at the timepoints 2.5, 3, 3.5, 4, 4.5, 5, > 5 to ≤ 10 and > 10



<Protocol: Janssen OZ1-HV1-101/102/202>


years post infusion will be presented. In addition Spearman's rank correlation co-efficient and its associated p-value overall timepoints will be presented. Similar presentations will be made for patients experiencing at least one NSRAEs.

#### 8.2.6. Summary of Patient Death

AEs where the outcome recorded as 'fatal' and/or seriousness is recorded as 'death' will be tabulated by system organ class and preferred term. Counts will be given for both system organ class and preferred term. Deaths will be identified within the relevant preferred term.

#### 8.3. PREDOMINANT INTEGRATION SITE TEST

Predominant integration site is defined as an integration site which has a density of at least 50% of the total signal detected by PCR, when the percentage of cells marked by the vector (quantitative OZ1/LNL6 DNA PCR) is greater than 1% of the test cell population. Results are recorded as part of the initial study information and at each follow-up visit.

A confirmed finding of a predominant integration site is a finding that is present on at least 2 consecutive samples. A predominant integration site finding will be reported as an SAE. Predominant integration site results will be listed only, no summary tables will be presented.

#### 8.4. CBC/DIFFERENTIAL AND PLATELETS

CBC/differential and platelets (haematocrit, red blood count, haemoglobin, white blood count, platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils) will be recorded as part of the initial study information and at each follow-up visit. CBC/differential and platelets data will be recorded in the units as pre-printed on the CRF. No conversion of these data to Standard International Units will be required.

CBC/differential and platelets values and change from baseline (2 years post infusion or nearest timepoint before starting long term follow-up) values will be summarized overall.

#### 8.5. CLINICAL HISTORY

Individual patient responses (Yes/No/Not Assessed) to the following questions will be recorded at 2.5 years post infusion and all subsequent follow-up visits:

Has the patient,

experienced new or exacerbated haematological disorders (including clinically significant laboratory abnormalities)?



<Protocol: Janssen OZ1-HV1-101/102/202>


had any new malignancies (including skin cancers)?

been exposed to possible therapeutic or environmental mutagenic agents?

experienced new or exacerbated pre-existing immunological/rheumatologic disorders?

experienced new or exacerbated pre-existing neurological disorders?

undergone a biopsy or surgical removal of a tumour?

For the last question, patient response to 'Was a sample collected for study assessment?' (Yes/No) will be recorded. If the response is 'Yes', the date of collection, will also be recorded. For the preceding questions, patient response to 'Is this possibly related to the gene transfer product will also be recorded?'.

The number and percentage of patients responding 'yes' to the above questions will be tabulated and presented by whether the information was received at a clinical visit, by telephone contact, and overall. The number of patients with clinical history information will also be presented. Percentages within each follow-up visit will be calculated using the number of patients with clinical history information at that visit.

#### 8.6. REPLICATION COMPETENT RETROVIRUS

Blood collected for PBMC archive will be used for Replication Competent Retrovirus (RCR) testing only if there is a clinically relevant AE, such as neoplasm, or an RCR test was positive, or not completed during the original study of the respective long term follow-up.

Positive findings will be analyzed further to confirm and identify any putative RCR. Any confirmed positive RCR finding will be reported as an SAE.

RCR results will be listed only. No summary tables will be presented.

#### 8.7. PHYSICAL EXAMINATION

A physical examination will be performed at each follow-up visit. Patient results (Not Done/Normal/Abnormal) and any description of an abnormal finding will be recorded for each body system (cardiovascular, respiratory, gastrointestinal, haematologic, endocrine, immunologic/rheumatologic, neurologic, dermatologic and other). Patient results will be listed only, no summary tables will be presented.

Research®

<Protocol: Janssen OZ1-HV1-101/102/202>


### 9. <u>INTERIM ANALYSES</u>

The first interim analysis of Year 5 follow-up data was done in 2011. The second interim analysis of Year 10 follow-up data has been done in 2016 followed by the final analysis expected in 2018.



<Protocol: Janssen OZ1-HV1-101/102/202>


# 10. CHANGES IN THE CONDUCT OF THE STUDY OR PLANNED ANALYSIS

#### 10.1. CHANGES IN THE CONDUCT OF THE STUDY

No changes are planned.

#### 10.2. CHANGES TO THE ANALYSES PLANNED IN THE STUDY

No changes to the analyses will be made.

Research®

<Protocol: Janssen OZ1-HV1-101/102/202>


### 11. REFERENCE LIST

N/A



<Protocol: Janssen OZ1-HV1-101/102/202>


### 12. PROGRAMMING CONVENTIONS

Listings will be sorted by long term follow-up study and patient identifier.

The dimensions and margins that will be used for the listings and table output produced via SAS are:

Paper: US letter

Pagesize: 43

Linesize: 132



<Protocol: Janssen OZ1-HV1-101/102/202>


### 13. <u>INDEX OF TABLES</u>

| Table Number | Table Description |
|---|---|
| 14.1.1 | Patient Disposition |
| | Including Reason for Discontinuation |
| | Summary Statistics: All Patients |
| 14.1.2 | Analysis Populations |
| | Summary Statistics: All Patients |
| 14.1.3 | Demographic Details |
| | Age, Gender and Race |
| | Summary Statistics: PP Population |
| 14.1.4 | Significant Medical History |
| | Time Since HIV-1 Infection |
| | Summary Statistics: PP Population |
| 14.1.5 | Treatment Details |
| | Summary Statistics: PP Population |
| 14.1.5a | Treatment Details (Study 202 only) |
| | Summary Statistics: PP Population |
| 14.1.6 | Compliance |
| | Visit Attendance |
| | Summary Statistics: PP Population |
| 14.2.1.1 | OZ1 and LNL6 DNA PCR |
| | Marking Parameters (PBMC) Over Time: Actual Values |
| | Summary Statistics: PP Population |
| 14.2.1.1a | OZ1 and LNL6 DNA PCR |
| | Marking Parameters (PBMC) Over Time: Actual Values (Study 202 only) |
| | Summary Statistics: PP Population |
| 14.2.1.2 | OZ1 and LNL6 DNA PCR |
| | Relationship of Marking Parameters (PBMC) with Calculated Dose, Age, Time on Study, |
| | Gender and Race |
| | Statistical Analysis: PP Population |
| 14.2.1.2a | OZ1 and LNL6 DNA PCR |
| | Relationship of Marking Parameters (PBMC) with Calculated Dose, Age, Time on Study, |
| | Gender and Race (Study 202 only) |
| | Statistical Analysis: PP Population |
| 14.3.1 | Overall Summary of Adverse Events |
| | Summary Statistics: Safety Population |
| 14.3.2 | Serious Adverse Events |
| | By System Organ Class, Preferred Term, Severity and Relationship including Patient ID |
| | Summary Statistics: Safety Population |
| 14.3.3 | Serious and Non Serious Related Adverse Events |
| | By System Organ Class, Preferred Term, Outcome and Relationship including Patient ID |
| | Summary Statistics: Safety Population |
| 14.3.4 | Time Adjusted Serious Adverse Events |
| | By System Organ Class and Preferred Term |
| | Summary Statistics: Safety Population |
| 14.3.5 | Serious and Non-Serious Related Adverse Events |
| | Relationship Between Time on Study and Related Serious and Non Serious Adverse |
| | Events |
| | Summary Statistics: Safety Population |



<Protocol: Janssen OZ1-HV1-101/102/202>


| 14.3.6 | Patient Death |
|---|---|
| | By System Organ Class and Preferred Term, Including Patient ID |
| | Summary Statistics: Safety Population |
| 14.4.1 | Clinical History |
| | Experienced new or exacerbated pre-existing haematological disorders |
| | (including clinically significant laboratory abnormalities)? |
| | Summary Statistics: PP Population |
| 14.4.2 | Clinical History |
| | Had any new malignancies (including skin cancers)? |
| | Summary Statistics: PP Population |
| 14.4.3 | Clinical History |
| | Been exposed to possible therapeutic or environmental mutagenic agents? |
| | Summary Statistics: PP Population |
| 14.4.4 | Clinical History |
| | Experienced new or exacerbated pre-existing immunologic/rheumatologic disorders? |
| | Summary Statistics: PP Population |
| 14.4.5 | Clinical History |
| | Experienced new or exacerbated pre-existing neurological disorders? |
| | Summary Statistics: PP Population |
| 14.4.6 | Clinical History |
| | Undergone a biopsy or surgical removal of a tumor? |
| | Summary Statistics: PP Population |
| 14.5.X | CBC/Differential and Platelets |
| | Parameter X |
| | Summary Statistics: PP Population |
| L | l |



<Protocol: Janssen OZ1-HV1-101/102/202>


### 14. <u>INDEX OF FIGURES</u>

| Figure Number | Figure Description |
|---------------|-------------------------------------------------------|
| 14.1.1 | OZ1 & LNL6 DNA PCR |
| | % of Patients Tested with a Detected Result Over Time |
| | By Study : PP Population |
| 14.1.2 | OZ1 & LNL6 DNA PCR |
| | % of Patients Tested with a Detected Result Over Time |
| | OZ1-HV1-102/202 : PP Population |
| 14.1.3 | OZ1 & LNL6 DNA PCR |
| | % of Patients Tested with a Detected Result Over Time |
| | OZ1-HV1-101/102/202 : PP Population |



<Protocol: Janssen OZ1-HV1-101/102/202>


### 15. <u>INDEX OF LISTINGS</u>

| Listing Number | Listing Description |
|----------------|------------------------------------------------|
| 16.2.1.1 | Discontinuation Details |
| | By Study and Patient |
| | All Patients |
| 16.2.1.2 | Patient Re-instatement Details |
| | By Study and Patient |
| 10010 | All Patients |
| 16.2.1.3 | Reason for Exclusion from Analysis Populations |
| | By Study and Patient All Patients |
| 16.2.2 | Demographic Details |
| 10.2.2 | By Study and Patient |
| | All Patients |
| 16.2.3 | Significant Medical History |
| 10.2.0 | By Study and Patient |
| | All Patients |
| 16.2.4 | Initial Study Information |
| | Treatment Details |
| | By Study and Patient |
| | All Patients |
| 16.2.5.1 | Compliance Visit Attendance |
| | By Study and Patient |
| | All Patients |
| 16.2.5.2.1 | PBMC Analysis Details |
| | OZ1 & LNL6 DNA PCR |
| | By Study and Patient All Patients |
| 16.2.5.2.2 | PBMC Analysis Details |
| 10.2.3.2.2 | OZ1 & LNL6 DNA PCR |
| | By Study and Patient |
| | Patients with Quantifiable Measurements |
| 16.2.5.2.3 | PBMC Analysis Details |
| | OZ1 RNA RT-PCR |
| | Study OZ1-HVI-202 |
| | All Patients |
| 16.2.5.2.4 | PBMC Analysis Details |
| | RCR |
| | By Study and Patient |
| | All Patients |
| 16.2.6 | Predominant Integration Site |
| | Marking >1% |
| | By Study and Patient All Patients |
| 16.2.7 | Integration Re-Test Details |
| 10.4.1 | By Study and Patient |
| | All Patients |
| 16.2.8.1 | Patient Death |
| | By Study and Patient |



<Protocol: Janssen OZ1-HV1-101/102/202>


| | All Deficete |
|---|---|
| | All Patients |
| 16.2.8.2 | Serious Adverse Events |
| | By Study and Patient |
| | All Patients |
| 16.2.8.3 | Non-Serious Related Adverse Events |
| | By Study and Patient |
| | All Patients |
| 16.2.9 | Central Laboratory Testing |
| | Blood Collection Details |
| | By Study and Patient |
| | All Patients |
| 16.2.10 | RCR Test Details |
| | By Study and Patient |
| | All Patients |
| 16.2.11 | CBC/Differential and Platelets |
| | By Study and Patient |
| | All Patients |
| 16.2.12 | Clinical History |
| | By Study and Patient |
| | All Patients |
| | (Pgm Note: Incorporate flag to determine whether data was collected at clinical visit or |
| | telephone contact) |
| 16.2.13 | Physical Examination |
| | By Study and Patient |
| | All Patients |



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.1.1

Page x of y

## Patient Disposition Including Reason for Discontinuation Summary Statistics: All Patients

OZ1-HV1-101 (N = X) n (%)

OZ1-HV1-102 (N = XX)n (%) OZ1-HV1-202 (N = XX) n (%)

Overall
(N = XX)
n (%)

Patients Ongoing (Never Discontinued)

Patients Discontinued (and Re-instated)
Reason
Patient request
Randomized to placebo arm in OTH/OZ1-INT-1
Lost to follow up
Regulatory authority request
Study termination
Other

Patients Discontinued (Never Re-instated)
Reason
Patient request
Randomized to placebo arm in OTH/OZ1-INT-1
Lost to follow up
Regulatory authority request
Study termination
Other

Note: Data summarized in this table are presented in data listing x.x It is possible that patients may withdraw on more than one occasion.

DDMMMYYY HH:MM

Prgm note: Percentage is based on N

Final SAP: 07Nov2017 CONFIDENTIAL




<Protocol: Janssen OZ1-HV1-101/102/202>

<INC code: 1003733>

<SAP Version: 3.0>

Janssen - OZ1-HVI-101/102/202

TABLE 14.1.2

Page x of y

#### Analysis Populations Summary Statistics: All Patients

| OZ1-HV1-101 | OZ1-HV1-102 | OZ1-HV1-202 | Overall |
|-------------|-------------|-------------|---------|
| (N = X) | (N = XX) | (N = XX) | (N=XX) |
| n (%) | n (%) | n (%) | n (%) |

Patients entered long term follow-up

Patients in safety population

Patients in per protocol population

Note: Data summarized in this table are presented in data listing x.x

DDMMMYYY HH:MM

Final SAP: 07Nov2017 


<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.1.3

Page x of y

Demographic Details
Age, Gender and Race
Summary Statistics: PP Population

| | | | OZ1-HV1-101 $(N = X)$ | OZ1-HV1-102<br>(N = XX) | OZ1-HV1-202 (N = XX) | Overall (N = XX) |
|---|---|---|---|---|---|---|
| Age(years) | At infusion | Mean<br>Median<br>SD<br>Min<br>Max<br>n | | | | |
| | At study start<br>(2 years post infusion) | Mean<br>Median<br>SD<br>Min<br>Max<br>n | | | | |
| | At database lock cut off | Mean<br>Median<br>SD<br>Min<br>Max<br>n | | | | |

Note: Data summarized in this table are presented in data listing x.x

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.1.3

Page x of y

# Demographic Details Age, Gender and Race Summary Statistics: PP Population

| | | | OZ1-HV1-101 $(N = X)$ | OZ1-HV1-102 $(N = XX)$ | OZ1-HV1-202<br>(N = XX) | Overall<br>(N = XX) |
|---|---|---|---|---|---|---|
| Gender | Male | n (%) | | | | |
| | Female | n (%) | | | | |
| Race | Aboriginal | n (%) | | | | |
| | African American | n (%) | | | | |
| | American Indian | n (%) | | | | |
| | Asian | n (%) | | | | |
| | Caucasian | n (%) | | | | |
| | Hispanic | n (%) | | | | |
| | Maori/Polynesian | n (%) | | | | |
| | Other | n (%) | | | | |

Note: Data summarized in this table are presented in data listing  $\mathbf{x}.\mathbf{x}$ 

Programming Note: Overall column will be populated for Race only

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.1.4

Page x of y

Significant Medical History Time Since HIV-1 Infection Summary Statistics: PP Population

| Time Since HIV-1 | OZ1-HV1-101 | OZ1-HV1-102 | OZ1-HV1-202 | Overall |
|-------------------|-------------|-------------|-------------|----------|
| Infection (years) | (N = X) | (N = XX) | (N = XX) | (N = XX) |

Mean Median SD Min Max

Note: Data summarized in this table are presented in data listing x.xTime since HIV-1 infection is derived as Year of diagnosis - (Date of Database lock + 1)

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.1.5

Page x of y

#### Treatment Details Summary Statistics: PP Population

| | | Cell | Туре |
|----------------------------------|--------|------|------|
| | | CD4 | CD34 |
| Time since infusion (years) | Mean | | |
| | Median | | |
| | SD | | |
| | Min | | |
| | Max | | |
| | n | | |
| Dose (x10 <sup>6</sup> cells/kg) | Mean | | |
| | Median | | |
| | SD | | |
| | Min | | |
| | Max | | |
| | n | | |
| Transduction efficiency | Mean | | |
| | Median | | |
| | SD | | |
| | Min | | |
| | Max | | |
| | n | | |
| Calculated dose (1) | Mean | | |
| | Median | | |
| | SD | | |
| | Min | | |
| | Max | | |
| | n | | |

Note: Data summarized in this table are presented in data listing x.x
(1) Calculated dose = Dose(CD4+ or CD34+)/(100 x transduction efficiency)
Programming note: Please repeat this table for 14.1.5a (Study 202 only)

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.1.6

Page x of y

# Compliance Visit Attendance Summary Statistics: PP Population

| Time since infusion | | OZ1-HV1-101 $(N = X)$ | OZ1-HV1-102 (N = XX) | OZ1-HV1-202 (N = XX) | Overall (N = XX) |
|---|---|---|---|---|---|
| ≤ 5yrs | Mean<br>Median<br>SD<br>Min<br>Max<br>n | | | | |
| > 5yrs ≤ 10yrs | Mean<br>Median<br>SD<br>Min<br>Max<br>n | | | | |
| Repeat for:<br>> 10yrs ≤ 15yrs<br>> 15 yrs | Mean<br>Median<br>SD<br>Min<br>Max<br>n | | | | |

Note: Data summarized in this table are presented in data listing x.x Compliance is calculated by (Number of Visit Eligible to Attend - Number of Visits Attended) / Number of Visit Eligible to Attend Repeat or unscheduled visits are not included in the above calculation.

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.2.1.1 Page x of y

OZ1 and LNL6 DNA PCR
Marking Parameters (PBMC)Over Time: Actual Values
Summary Statistics: PP Population

| | | | OZ1-HV1-102 / | |
|---|---|---|---|---|
| | | | OZ1-HV1-202 | Overall |
| Visit | Result | | (N = XX) | (N = XX) |
| 2 years post infusion | Analysed Sample | n | | |
| | Not Detected | n (%) | | |
| | 1/3 Detected * | n (%) | | |
| | 2/3 Detected * | n (%) | | |
| | 3/3 Detected * | n (%) | | |
| | Quantifiable OZ1 & LNL6 DNA Detected | n (%) | | |
| 2.5 years post infusion | Analysed Sample | n | | |
| | Not Detected | n (%) | | |
| | 1/3 Detected * | n (%) | | |
| | 2/3 Detected * | n (%) | | |
| | 3/3 Detected * | n (%) | | |
| | Quantifiable OZ1 & LNL6 DNA Detected | n (%) | | |
| 3 years post infusion | Analysed Sample | n | | |
| | Not Detected | n (%) | | |
| | Etc | | | |

Note: Data summarized in this table are presented in data listing  $\mathbf{x}.\mathbf{x}$ 

 ${\it DDMMMYYYY} \qquad {\it HH:MM}$ 

Prgm note: % based on N  $\,$ 

Programming note: Please repeat this table for 14.2.1.1a (Study 202 only)

<sup>\* =</sup> OZ1 & LNL6 DNA Detected but below the lower quantitative limit of the assay: 1/3 = 1 of the 3 triplicates of the sample were detected; 2/3 = 2 of the 3 triplicates of the sample were detected.



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.2.1.2 Page x of y

OZ1 and LNL6 DNA PCR

Relationship Between Marking Parameters (PBMC) and Calculated Dose, Age, Time on Study, Gender and Race Summary Statistics: PP Population

| | | | OZ1-HV1-102 / | |
|---|---|---|---|---|
| | | | OZ1-HV1-202 | Overall |
| Visit | PBMC versus | Statistic | (N = XX) | (N = XX) |
| 2 years post infusion | Calculated Dose | N (1)<br>Rho (2)<br>p-value | | |
| | Age (3) | N (1)<br>Rho (2)<br>p-value | | |
| | Time on Study | N (1)<br>Rho (2)<br>p-value | | |
| | Gender | N (1)<br>Chi-Square (4)<br>p-value | | |
| | Race (5) | N (1)<br>Chi-Square (4)<br>p-value | | |
| 2.5 years post infusion Etc | Calculated Dose | N (1)<br>Rho (2)<br>Etc | | |

Note: Data summarized in this table are presented in data listing x.x

- (1) N = number of patients with quantifiable OZ1 & LNL6 DNA detected
- (2) Rho = Spearman's Rank Correlation co-efficient
- (3) = Age at infusion



<Protocol: Janssen OZ1-HV1-101/102/202>


(4) = Chi-Square statistic

(5) = Race categories (Aboriginal, African American, American Indian, Asian, Caucasian, Hispanic, Maori/Polynesian, Other DDMMMYYYY HH:MM

Prgm note: Fishers Exact test may be presented if Chi-Square test is not appropriate Programming note: Please repeat this table for 14.2.1.2a (Study 202 only)



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.3.1


Overall Summary of Adverse Events Summary Statistics: Safety Population

| | OZ1-HV1-101<br>(N=xx) | OZ1-HV1-102<br>(N=xx) | OZ1-HV1-202<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| Number (%) of patients with at least one SAE | (2. 3337) | (2. 2227) | (21 2222) | (= |
| Number (%) of patients with at least one related SAE Number (%) of patients with at least one severe related SAE Number (%) of patients with least one NSRAE Number (%) of patients with SAE/NSRAE leading to death | | | | |
| Number of SAEs Number of related SAEs | | | | |
| Number of severe related SAEs<br>Number of NSRAEs<br>Number of SAE/NSRAE leading to death | | | | |

Note: Data summarized in this table are presented in data listing x.x

SAE = Serious Adverse Event; NSRAE = Non-serious related adverse event

Drug-related adverse events are those events with a relationship of possible, probable or very likely

Events with missing severity are assumed to be the severe category

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.3.2


Serious Adverse Events
By System Organ Class, Preferred Term, Severity and Relationship including Patient ID
Summary Statistics: Safety Population

| | | | | | | OZ1-H | V1-101 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | | | | (N= | exx) | | | | | |
| Preferred Term | | Mild | | | Moderate | · | | Severe- | | Overall | | |
| | n (%) | NR | Rel | n (%) | NR | Rel | n (%) | NR | Rel | n (%) | NR | Rel |
| SYSTEM ORGAN CLASS 1 | 3 (x.x) | 1 | 2 | 0 | 0 | 0 | 1 (x.x) | 0 | 1 | 4 (x.x) | 1 | 3 |
| PREFERRED TERM 1 | 1 (x.x) | 1<br>R0001 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (x.x) | 1 | 0 |
| PREFERRED TERM 2 | 1 (x.x) | 0 | 1<br>R0002 | 0 | 0 | 0 | 1 (x.x) | 0 | 1<br>R0004 | 2 (x.x) | 0 | 2 |
| PREFERRED TERM 3 | 1 (x.x) | 0 | 1<br>R0003 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (x.x) | 0 | 1 |
| SYSTEM ORGAN CLASS A<br>PREFERRED TERM 1<br>PREFERRED TERM 2 | | | | | | | | | | | | |
| ETC | | | | | | | | | | | | |

Note: Data summarized in this table are presented in data listing x.x

NR = Not related (those events with a relationship of not related or doubtful

Rel = Drug-related adverse events (those events with a relationship of possible, probable or very likely)

Events with missing severity are assumed to be the severe category

DDMMMYYYY HH:MMM

Prgm note: This table will continue for OZ1-HV1-102, OZ1-HV1-202 and Overall

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.3.3


Serious and Non-Serious Related Adverse Events
By System Organ Class, Preferred Term, Outcome and Relationship including Patient ID
Summary Statistics: Safety Population

| | | | | | | OZ | 1-HV1-101 | 5. | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| System Organ Class | | | | | | | (N=xx) | | | | | |
| Preferred Term | Recov | ered\Reso | lved | Recove | ring\Re | solving | Not Rec | overed\N | ot Resolved | Recover | ed with | n sequelea |
| | n (%) | NR | Rel | n (%) | NR | Rel | n (%) | NR | Rel | n (%) | NR | Rel |
| SYSTEM ORGAN CLASS 1 | 3 (x.x) | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 4 (x.x) | 1 | 3 |
| | | | | | | | (x.x) | | | | | |
| PREFERRED TERM 1 | 1 (x.x) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (x.x) | 1 | 0 |
| | | R0001 | | | | | | | | | | |
| PREFERRED TERM 2 | 1 (x.x) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 (x.x) | 0 | 2 |
| | | | | | | | (x.x) | | | | | |
| | | | R0002 | | | | | | R0004 | | | R0005<br>R0006 |
| PREFERRED TERM 3 | 1 (x.x) | 0 | 1<br>R0003 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (x.x) | 0 | 1 |

SYSTEM ORGAN CLASS A
PREFERRED TERM 1
PREFERRED TERM 2

ETC

Note: Data summarized in this table are presented in data listing X.X.X.X

NR = Not related (those events with a relationship of not related or doubtful

Rel = Drug-related adverse events (those events with a relationship of possible, probable or very likely)

DDMMMYYYY HH:MMM

Prgm note: This table will continue for Fatal and Unknown categories and for OZ1-HV1-102, OZ1-HV1-202 and Overall

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.3.4


Time Adjusted Serious Adverse Events By System Organ Class, Preferred Term Summary Statistics: Safety Population

System Organ Class

Preferred Term OZ1-HV1-101 OZ1-HV1-102

OZ1-HV1-202

Overall

SYSTEM ORGAN CLASS 1 Number of events Event rate per year PREFERRED TERM 1 Number of events Event rate per year PREFERRED TERM 2 Number of events Event rate per year SYSTEM ORGAN CLASS 2 Number of events Event rate per year PREFERRED TERM 1

Number of events Event rate per year ETC

Note: Data summarized in this table are presented in data listing X.X.X.X

Event rate per year = Number of related SAEs / Patient years in long term follow-up

DDMMMYYYY HH:MMM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.3.5


Serious and Non-Serious Related Adverse Events Relationship Between Time on Study and Related Serious and Non Serious Adverse Events Summary Statistics: Safety Population

| | | | OZ1-HV1-102 / | |
|---|---|---|---|---|
| Visit | | Statistic | OZ1-HV1-202 $(N = XX)$ | Overall (N = XX) |
| 2.5 years post infusion | SAE | N (1)<br>Rho (2)<br>p-value | | |
| | NSRAE | N (1)<br>Rho (2)<br>p-value | | |
| 3 years post infusion | SAE | N (1)<br>Rho (2)<br>p-value | | |
| | NSRAE | N (1)<br>Rho (2)<br>p-value | | |
| 3.5 years post infusion | N (1)<br>Rho (2)<br>p-value | SAE | | |
| Etc | Etc | Etc | | |

Note: Data summarized in this table are presented in data listing x.x

- (1)  $\ensuremath{\mathtt{N}}$  = number of patients experiencing at least one event
- (2) Rho = Spearman's Rank Correlation co-efficient

DDMMMYYYY HH:MMM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.3.6


Patient Death

By System Organ Class, Preferred Term including Patient ID

Summary Statistics: Safety Population

| System Organ Class<br>Preferred Term | OZ1-HV1-101<br>(N=xx) | OZ1-HV1-102<br>(N=xx) | OZ1-HV1-202<br>(N=xx) | Overall (N=xx) |
|---|---|---|---|---|
| SYSTEM ORGAN CLASS 1 | 2 | 1 | 2 | 5 |
| PREFERRED TERM 1 | 1<br>R0001 | 1<br>R0002 | 1<br>R0003 | 3 |
| PREFERRED TERM 2 | 1<br>R0004 | 0 | 1<br>R0005 | 2 |
| SYSTEM ORGAN CLASS 2 | 1 | 0 | 0 | 1 |
| PREFERRED TERM 1 | 1<br>R0004 | 0 | 0 | 1 |
| PREFERRED TERM 2<br>ETC | etc | | | |

Note: Data summarized in this table are presented in data listing X.X.X.X Death is defined as an AE outcome recorded as fatal and/or a AE seriousness recorded as death

DDMMMYYYY HH:MMM

Suggest add footnote to define how these are selected (AEs with outcome='fatal')?

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202

TABLE 14.4.1


Clinical History

Experienced new or exacerbated pre-existing haematological disorders (including clinically significant laboratory abnormalities)?

Summary Statistics: PP Population

| | | Telephone | | |
|---|---|---|---|---|
| | | Clinical Visit | Contact | Overall |
| | | (N = XX) | (N = XX) | (N = XX) |
| Long Term Follow-up Visit | Response | n (%) | n (%) | n (%) |
| 0.5 | 3.7* | | | |
| 2.5 yrs post infusion | $N^*$ | | | |
| | Yes | | | |
| | Related | | | |
| | Not Related | | | |
| | No | | | |
| | Not Assessed | | | |
| 3 yrs post infusion | $N^*$ | | | |
| | Yes | | | |
| | Related | | | |
| | Not Related | | | |
| | No | | | |
| | Not Assessed | | | |
| 3.5 yrs post infusion | $N^{\star}$ | | | |
| Etc | Etc | | | |

Note: Data summarized in this table are presented in data listing X.X.X.X  $N^*$  represents the number of patients responding at each visit and is used as the denominator to calculate percentage DDMMYYYYY HH:MM

Similar tables will appear for:
Had any new malignancies (including skin cancers)?
Been exposed to possible therapeutic or environmental mutagenic agents?
Experienced new or exacerbated pre-existing immunologic/rheumatologic disorders?

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Experienced new or exacerbated pre-existing neurological disorders? Undergone a biopsy or surgical removal of a tumor?



<Protocol: Janssen OZ1-HV1-101/102/202>


Janssen - OZ1-HVI-101/102/202 TABLE 14.5.X Page x of y

# CBC/Differential and Platelets $Parameter\ (units)$ Summary Statistics: PP Population

Overall Post infusion ----- Result ---------- Change from Baseline -----Visit std median min max n mean std median min max n 2 years 2.5 years 3 years 3.5 years 4 years 4.5 years 5 years Etc...

Note: Data summarized in this table are presented in data listing x.x

Baseline is the 2 year post infusion visit or nearest timepoint before start of long term follow-up

DDMMMYYYY HH:MM

Final SAP: 07Nov2017 



<Protocol: Janssen OZ1-HV1-101/102/202>


Below is an example of a typical listing ie Protocol, Treatment, Dose and Patient ID will appear on all listings. For some lisitings this may mean that space is restricted for other data and the listing may be split over more than one page.

Data Listing 16.2.X Listing Description All Patients

| Protocol | Treatment | Dose | Patient ID | Listed data1 | Listed data2 | Listed data3 | Listed data4 |
|---|---|---|---|---|---|---|---|
| <i>ie</i> OZ1-HIV-1- | OZI | CD4 or | | | | | |
| or OZ1-HIV-1-<br>102 | or LNL6 | CD34 | | | | | |
| or OZ1-HIV-1-<br>202 | or OZ1&LNL6 | | | | | | |
| | or placebo | | | | | | |